CLINICAL TRIAL: NCT03052569
Title: Expanded Access to RXDX-105 for the Treatment of Cancers With RET Alterations
Brief Title: Expanded Access to RXDX-105 for Cancers With RET Alterations
Status: No longer available | Type: Expanded Access
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: RXDX-105 - EAP
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Cancers With RET Alterations
MeSH Terms: interventions — agerafenib

INTERVENTIONS:
Drug: RXDX-105 — Oral Capsules

SUMMARY:
Expanded access to RXDX-105 will be given to patients with cancers harboring RET alterations who have not received TKIs that target RET alterations, who do not qualify for participation in, or who are otherwise unable to access, an ongoing clinical trial for RXDX-105.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced cancer with RET alterations
* Unable to participate in an ongoing RXDX-105 clinical trial
* Willing and able to provide written, signed informed consent
* Medically suitable for treatment with RXDX-105

Exclusion Criteria:

* Prior treatment with a TKI that has activity against RET alterations
* Currently enrolled in an ongoing clinical study with any other investigational agent

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Www.Ignyta.Com, San Diego, California, United States